CLINICAL TRIAL: NCT07150559
Title: Arch-Clamping Technique Under Mild Hypothermia in Treating With Acute Type A Aortic Dissection: Study Protocol for a Multicenter, Three-arm, Open-label, Randomized, Parallel-controlled Trial
Brief Title: Arch-Clamping Technique Under Mild Hypothermia in Treating With Acute Type A Aortic Dissection
Acronym: AHEAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Yan'an Affiliated Hospital of Kunming Medical University (Other); Xiangya Hospital of Central South University (Other); West China Hospital (Other); Guangzhou First People's Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Xijing Hospital，FMMU (Unknown)
Responsible Party: Principal Investigator, Junming Zhu, Vice Chairman, Aortic Surgery Committee of Chinese Association of Cardiovascular Surgeons; President, Beijing Society for Thoracic and Cardiovascular Surgery; Director, Center for Aortic Surgery, Beijing Anzhen Hospital, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023ZD0504402
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-09

CONDITIONS: Acute Type A Aortic Dissection; Hypothermia; Total Aortic Arch Replacement; Frozen Elephant Trunk; Bilateral Antegrade Cerebral Perfusion
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, three-arm, open-label, randomized, parallel-controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arch-clamping under mild hypothermia (Experimental): TAR + FET procedure is performed using arch-clamping technique under mild hypothermia.
  Interventions: Procedure: Arch-Clamping Technique under Mild Hypothermia
- Arch-clamping under moderate hypothermia (Experimental): TAR + FET procedure is performed using arch-clamping technique under moderate hypothermia.
  Interventions: Procedure: Arch-Clamping Technique under Moderate Hypothermia
- Sun's procedure using bACP (Active Comparator): Total arch replacement and frozen elephant trunk implantation with moderate hypothermic circulatory arrest.
  Interventions: Procedure: Total Arch Replacement combined Frozen Elephant Trunk Implantation using Bilateral Antegrade Cerebral Perfusion under Moderate Hypothermic Circulatory Arrest

INTERVENTIONS:
Procedure: Arch-Clamping Technique under Mild Hypothermia — This procedure is performed under mild hypothermia. The branch arteries of the arch are reconstructed using the side arms of a Y-shaped graft, which allows bilateral antegrade cerebral perfusion (bACP) through the right axillary artery. A FET is deployed in the descending aorta and clamped together with the autologous aorta immediately, then distal perfusion is restored through the femoral artery. After the proximal procedures are completed, the distal anastomosis is performed in an end-to-end fashion. Finally, the main trunk of the Y-shaped graft is anastomosed to the proximal grafts.
  Arms: Arch-clamping under mild hypothermia
Procedure: Arch-Clamping Technique under Moderate Hypothermia — This procedure is performed under moderate hypothermia. The branch arteries of the arch are reconstructed using the side arms of a Y-shaped graft, which allow bACP through the right axillary artery. A FET is deployed in the descending aorta and clamped together with the autologous aorta immediately, then distal perfusion is restored through the femoral artery. After the proximal procedures are completed, the distal anastomosis is performed in an end-to-end fashion. Finally, the main trunk of the Y-shaped graft is anastomosed to the proximal grafts.
  Arms: Arch-clamping under moderate hypothermia
Procedure: Total Arch Replacement combined Frozen Elephant Trunk Implantation using Bilateral Antegrade Cerebral Perfusion under Moderate Hypothermic Circulatory Arrest — This procedure is performed using bACP under MHCA, which involves FET deployment in the descending aorta followed by total arch replacement with a four-branched vascular graft. Deployment of the FET and suture of the distal anastomosis are completed during bACP. MHCA is terminated and distal reperfusion is initiated once the distal anastomosis is completed, and the left carotid artery is reconstructed first (after which bACP is stopped, rewarming is started and the brain is perfused bilaterally). The root or valve procedures and some concomitant operations, if indicated, are performed during the cooling phase.
  Arms: Sun's procedure using bACP

SUMMARY:
The study is a multicenter, three-arm, open-label, randomized, parallel-controlled trial, which plans to enroll 306 participants diagnosed with acute type A aortic dissection (ATAAD) from 7 hospitals in China. All patients receive total arch replacement (TAR) combined with frozen elephant trunk (FET) implantation and are randomized to Group 1 (arch-clamping technique under mild hypothermia), Group 2 (arch-clamping technique under moderate hypothermia) and Group 3 (Sun's procedure using bilateral antegrade cerebral perfusion) in the ratio of 1:1:1. After a 1-year follow-up, the validity and safety of the mild hypothermic arch-clamping technique for ATAAD was evaluated via the incidence of major adverse events including death, renal replacement therapy, stroke, and paraplegia, as well as times of circulatory arrest, cardiopulmonary bypass, and mechanical ventilation, and length of ICU stay.

ELIGIBILITY:
Inclusion Criteria:

1. Aortic CTA confirmed as ATAAD according to the 2022 ACC/AHA Guideline for the Diagnosis and Management of Aortic Disease;
2. Adult patients (18-70 years) weighing 50-120 kg;
3. Time interval between the onset of symptoms and operation is less than 14 days;
4. Indications for total aortic arch replacement are available;
5. Signed informed consent and availability for follow-up.

Exclusion Criteria:

1. History of chronic renal failure, hepatocirrhosis, and hepatic insufficiency;
2. Severe gastrointestinal complications of non-aortic dissection, such as mesenteric ischemia, gastrointestinal bleeding, hepatopancreaticobiliary dysfunction, and intestinal obstruction;
3. History of severe cerebral infarction (with cerebral infarction sequels);
4. Preoperative intubation or unconsciousness;
5. Inflammatory aortic diseases, such as Takayasu arteritis and Behçet's disease, etc;
6. History of infectious aortic diseases;
7. History of cardiac and aortic surgery;
8. History of malignancy or previous radiotherapy;
9. Pregnant or feeding women, or anyone planning to reproduce during the test period;
10. Without an informed consent signature;
11. Participating in any other clinical trial;
12. Having other causes not eligible for operation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Major adverse events | Thirty days and 12 months after the operation
  Major adverse events include death, renal replacement therapy, stroke, and paraplegia

SECONDARY OUTCOMES:
Circulatory arrest time | During surgery
  Time interval between ceasing and restarting cardiopulmonary bypass when core temperature reaches moderate hypothermia.
Cardiopulmonary bypass time | During surgery
  Start-to-end time of cardiopulmonary bypass to complete aortic repair.
Mechanical ventilation time | Discharge / 30 days after operation
  Time interval between mechanical ventilation and extubation after operation
The length of ICU stay | Discharge / 30 days after operation
  Time interval from ICU admission to transfer or death

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No